CLINICAL TRIAL: NCT04420325
Title: COronary and MICrocirculatory Measurements in Patients With Aortic Valve, the COMIC AS Study.
Brief Title: COronary and MICrocirculatory Measurements in Patients With Aortic Valve Stenosis.
Acronym: COMIC-AS
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: AZ Delta (Other); University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Other Study IDs: S63740
Record Dates: First submitted 2020-06-03; First posted 2020-06-09 (Actual); Results first posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-06

CONDITIONS: Aortic Stenosis; Coronary Artery Disease
MeSH Terms: conditions — Aortic Valve Stenosis; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Before IMR measurement, a peripheral blood sample (10cc EDTA, citrate and 2.5mL PaxGene® RNA tube) will be obtained to assess platelet function and for biomarker evaluation (RNA analysis).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Although concomitant coronary artery disease (CAD) is frequent in patients with severe aortic stenosis (AS), hemodynamic assessment of CAD severity in patients undergoing valve replacement for severe AS is challenging. Myocardial hypertrophic remodeling interferes with coronary blood flow and may influence the values of fractional flow reserve (FFR) and nonhyperemic pressure ratios (NHPRs). The aim of the current study is to investigate the effect of the AS and its treatment on current indices used for evaluation of CAD. The investigators will compare intracoronary hemodynamics before, immediately after, and 6 mo after aortic valve replacement (AVR) when it is expected that microvascular function has improved. Furthermore, the investigators will compare FFR and resting full-cycle ratio (RFR) with myocardial perfusion single-photon emission-computed tomography (SPECT) as indicators of myocardial ischemia in patients with AS and CAD. One-hundred consecutive patients with AS and intermediate CAD will be prospectively included. Patients will undergo pre-AVR SPECT and intracoronary hemodynamic assessment at baseline, immediately after valve replacement [if transcatheter AVR (TAVR) is chosen], and 6 mo after AVR. The primary end point is the change in FFR 6 mo after AVR. Secondary end points include the acute change of FFR after TAVR, the diagnostic accuracy of FFR versus RFR compared with SPECT for the assessment of ischemia, changes in microvascular function as assessed by the index of microcirculatory resistance (IMR), and the effect of these changes on FFR. The present study will evaluate intracoronary hemodynamic parameters before, immediately after, and 6 mo after AVR in patients with AS and intermediate coronary stenosis. The understanding of the impact of AVR on the assessment of FFR, NHPR, and microvascular function may help guide the need for revascularization in patients with AS and CAD planned for AVR.

DETAILED DESCRIPTION:
https://journals.physiology.org/doi/full/10.1152/ajpheart.00541.2021?rfr_dat=cr_pub++0pubmed&url_ver=Z39.88-2003&rfr_id=ori%3Arid%3Acrossref.org

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient undergoing the procedure is older than 18 years, has severe aortic valve stenosis (according to ESC guidelines) and is planned for cardiac catheterization as part of the pre-operative (SAVR) or pre-percutaneous (TAVI) work up.

  2. The patient has an intermediate (50-90%) coronary lesion that requires further evaluation.

  3. The patient undergoing the procedure is male, or if female, has no childbearing potential or is not pregnant.

Exclusion Criteria:

1. The procedure is an emergency and/or the patient is unstable.
2. Pregnancy or lactation
3. Haemodynamically unstable patients
4. Killip class III-IV heart failure
5. Previous coronary artery by-pass in the artery being assessed
6. Contra-indications for adenosine administration: severe asthma or pre-existing type 2 AV-block
7. No significant coronary artery disease (<50% stenosis on angiography).
8. Critical coronary artery disease deemed by the Heart Team to require immediate revascularization
9. Patients will be excluded from the SPECT study (secondary objective) if they have a left main coronary stenosis >50%, triple vessel disease, previous myocardial infarction in the same coronary artery & tandem lesions (separated by >10mm) requiring independent evaluation in the same coronary artery since these factors interfere with the SPECT analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing routine cardiac catheterization during preparation for TAVI or SAVR, who are found to have coronary artery disease, will be approached to take part.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Dubois, MD, PhD, Principal Investigator — UZ Leuven
Locations (3):
- Belgium (3):
  - UZ Leuven, Leuven, Vlaams-brabant
  - University hospital Antwerp, Antwerp
  - AZ Delta, Roeselare

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Rationale and Design paper — https://pubmed.ncbi.nlm.nih.gov/34676781/

RESULTS

PARTICIPANT FLOW:
Groups:
- Entire Study Population: Patients with AS undergoing TAVI or SAVR
Period: Overall Study
Arm/Group | Entire Study Population
Started | 116
Completed | 84
Not Completed | 32

BASELINE CHARACTERISTICS:
Population: Entire study population
Arm/Group | Entire Study Population
Number analyzed (Participants) | 116
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.48 (8.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 69
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 116
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 116

OUTCOME MEASURES:

1. Primary Outcome: FFR 6 Months After SAVR/TAVI.
Description: Aortic valve intervention can potentially result in a change in fractional flow reserve (FFR) 6 months after SAVR/TAVI.
  FFR is the ratio of two intra-coronary measurements (Distal coronary pressure divided by proximal coronary pressure) and can range from 0.0-1.0.
  A lower FFR means that the lesion is more severe and therefore a higher FFR is considered better. The threshold to speak about hemodynamic significant of a lesion is 0.80. If the lesion has an FFR of ≤ 0.80 means the lesions is significant and treatment is necessary.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Entire Study Population
Number analyzed (Participants) | 116
ratio | -0.0279 (0.0368)

2. Secondary Outcome: IMR 6 Months After SAVR/TAVI.
Description: Measurement of IMR in patients with AS prior to intervention and 6 months after TAVI/SAVR.
  IMR is unitless and gives a description of coronary microvascular resistance, it can range from 0-100.
  Lower values are considered better as they are related with better microvascular function and health.
  If the IMR > 25 we say microvascular dysfunction is present and treatment is considered necessary.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Unitless
Arm/Group | Entire Study Population
Number analyzed (Participants) | 116
Unitless | -2.8150 (12.1600)

3. Secondary Outcome: FFR Versus RFR to Determine Ischemia.
Description: Comparison of the diagnostic performance of FFR versus RFR compared with SPECT ischemia.
  The higher the Area under the curve the better. The range is 0.0-1.0. An area under the curve for a ROC model is considered excellent if > 0.8.
Time Frame: Baseline
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Entire Study Population
Number analyzed (Participants) | 116
probability | 0.8719 [0.8040 to 0.9397]

ADVERSE EVENTS:
Time Frame: From inclusion to 6 months
Arm/Group | Entire Study Population
All-Cause Mortality (participants affected / at risk) | 0/116
Serious Adverse Events (participants affected / at risk) | 0/116
Other Adverse Events (participants affected / at risk) | 0/116

LIMITATIONS AND CAVEATS:
First, microvascular function analysis was based on bolus-thermodilution,recent studies have shown that continuous coronary thermodilution may have better reproducibility. Second, myocardial perfusion SPECT is not the gold standard for non-invasive detection of ischemia.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT04420325/Prot_SAP_000.pdf